CLINICAL TRIAL: NCT05707091
Title: Effects of Low Laser Therapy on Facial Motor Functions Function and Synkinesis in Patients With Bell's Palsy
Brief Title: Low Laser Therapy on Facial Motor Functions Function and Synkinesis in Patients With Bell's Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0216
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Bell's Palsy
MeSH Terms: conditions — Bell Palsy | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level laser therapy (Experimental): Patients assigned to experimental group received low level laser therapy and conventional therapy. Treatment frequency was five sessions/week for 4 weeks. . For laser therapy, Omega laser system used with infrared probes of 830 nm wavelength and 100 mW output power, average energy density of 10 J/cm2 , frequency of 1 KHz, and a duty cycle of 80 % in one group. In all cases, the laser was in direct contact with the superficial roots of the facial nerve on the affected side. And was applied for 2 min and 5 s per point for 8 points.
  Interventions: Other: Low level laser therapy and conventional therapy
- Conventional therapy (Experimental): Group B was treated with conventional therapy. The interrupted galvanic electrical impulses with the duration of 3-30 milliseconds, the tolerable intensity was applied over the motor points of each facial muscle. A total of 30-60 electrical twitch induced muscle contractions will be maintained for each muscle. The facial muscles exercise training with mirror-visual feedback was progressed to resisted exercises by self and/or therapist-assistance. All exercises were demonstrated to participants by the therapist's efforts and instructed the participants to continue the exercises twice a day for 10-15 minutes. A pictorial leaflet of facial expressions exercises with appropriate instructions to perform exercises. Treatment frequency was five sessions/week for 4 weeks.
  Interventions: Procedure: Conventional therapy

INTERVENTIONS:
Other: Low level laser therapy and conventional therapy — One group treated with low level laser therapy along with conventional therapy
  Arms: Low level laser therapy
Procedure: Conventional therapy — Group B treated with ems and exercises
  Arms: Conventional therapy

SUMMARY:
To determine the effects of low-level laser therapy on facial motor functions and synkinesis in patients with bell's palsy

DETAILED DESCRIPTION:
A randomised controlled trial tested low-level laser therapy (LLLT) for bell's palsy. Lahore's Ittefaq Hospital selected 32 bell's palsy patients for the research. The Facial Disability Index (FDI), House-Brackmann Scale (HBS), and Sunnybrook Facial Grading System were used to collect data over ten months (SFG). LLLT and conventional therapy were randomly assigned to two groups. SPSS 25 compared pre- and post-treatment values of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Male female diagnosed with idiopathic Bell's palsy by physician
* age 30-60years
* Bell's palsy in patients having known history of hypertension
* Bell's palsy in patients having known history of diabetes

Exclusion Criteria:

* Participants with a middle ear infection
* parotid gland tumor
* malignant otitis external
* Tumors in the base of the lateral skull
* upper motor neuron facial palsy
* segmental muscle weakness
* and recurrent episodes of facial paralysis, polyneuropathies

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Facial disability index | 4 weeks
  To access the physical well-being
Housebrackmann scale | 4 weeks
  To grade the facial muscle weakness
Sunnybrook facial grading | 4 weeks
  To acess symmetry and synkinesis

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MsOmpt, Principal Investigator — Riphah International University
Locations (1):
- Ali raza, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aghamohamdi D, Fakhari S, Farhoudi M, Farzin H. The Efficacy of Low-Level Laser Therapy in the Treatment of Bell's Palsy in Diabetic Patients. J Lasers Med Sci. 2020 Summer;11(3):310-315. doi: 10.34172/jlms.2020.52. Epub 2020 Jun 21. PMID 32802293
- [Background] Ordahan B, Karahan AY. Role of low-level laser therapy added to facial expression exercises in patients with idiopathic facial (Bell's) palsy. Lasers Med Sci. 2017 May;32(4):931-936. doi: 10.1007/s10103-017-2195-9. Epub 2017 Mar 23. PMID 28337563
- [Background] de Oliveira RF, da Silva AC, Simoes A, Youssef MN, de Freitas PM. Laser Therapy in the Treatment of Paresthesia: A Retrospective Study of 125 Clinical Cases. Photomed Laser Surg. 2015 Aug;33(8):415-23. doi: 10.1089/pho.2015.3888. PMID 26226172
- [Background] Alayat MS, Elsodany AM, El Fiky AA. Efficacy of high and low level laser therapy in the treatment of Bell's palsy: a randomized double blind placebo-controlled trial. Lasers Med Sci. 2014 Jan;29(1):335-42. doi: 10.1007/s10103-013-1352-z. Epub 2013 May 26. PMID 23709010
- [Background] Bylund N, Hultcrantz M, Jonsson L, Marsk E. Quality of Life in Bell's Palsy: Correlation with Sunnybrook and House-Brackmann Over Time. Laryngoscope. 2021 Feb;131(2):E612-E618. doi: 10.1002/lary.28751. Epub 2020 May 28. PMID 32463963